CLINICAL TRIAL: NCT02076152
Title: A Study to Evaluate Vascular Normalization in Patients With Recurrent Glioblastoma Treated With Bevacizumab Using FMISO PET and Vascular MRI
Brief Title: FMISO PET Study of Glioblastoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elizabeth R. Gerstner, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-482; R01CA129371 (NIH)
Record Dates: First submitted 2014-02-06; First posted 2014-03-03 (Estimated); Results first posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Recurrent Glioblastoma
Keywords: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab; Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FMISO PET & MRI Group 1 (Experimental): * Bevacizumab:
    -- Bevacizumab will be administered at a dose of 10 mg/kg i.v. every 14 days per standard of care and the drug label. A cycle is defined as 28 days (1 month).
  * FMISO PET Scan
    * FMISO will be intravenously injected at a dose of 3.7 MBq/kg (0.1 mCi/kg) (maximum 260 MBq, 7 mCi) in < 15 mL. The IV will remain in place for injection of the gadolinium for the MRI scan. There will be one injection of FMISO in the PET protocol. Approximately 90 minutes after the injection, the PET scan will begin.
    * The PET scan will be approximately 60-75 minutes.
  * MRI -- Each MRI will last 60-75 minutes versus 45 minutes for standard brain MRIs.
  Interventions: Device: FMISO PET; Device: MRI; Drug: Bevacizumab
- FMISO PET & MRI Group 2 (Experimental): Bevacizumab + CCNU:
  * Bevacizumab will be administered at a dose of 10 mg/kg i.v. every 14 days per standard of care and the drug label. A cycle is defined as 28 days (1 month).
  * CCNU will be administered at a dose of 110 mg/m2 every 42 days per standard of care and the drug label. A cycle is defined as 28 days (1 month).
    -FMISO PET Scan
  * FMISO will be intravenously injected at a dose of 3.7 MBq/kg (0.1 mCi/kg) (maximum 260 MBq, 7 mCi) in < 15 mL. The IV will remain in place for injection of the gadolinium for the MRI scan. There will be one injection of FMISO in the PET protocol. Approximately 90 minutes after the injection, the PET scan will begin.
  * The PET scan will be approximately 60-75 minutes.
    - MRI
  * Each MRI will last 60-75 minutes versus 45 minutes for standard brain MRIs.
  Interventions: Device: FMISO PET; Device: MRI; Drug: Bevacizumab; Drug: CCNU

INTERVENTIONS:
Device: FMISO PET
Device: MRI — MR scans will be performed with the same sequences and in the same order during each visit, including T1- and T2-weighted volumetric images, fluid attenuated inversion recovery (FLAIR), contrast agent enhanced T1-weighted permeability, diffusion tensor imaging (DTI), T2/T2*-weighted perfusion scans, and MR Spectroscopy. The "Autoalign" package available from the manufacturer will be used to achieve the same slice prescription in the same patient at each visit. Each MRI will last 60-75 minutes versus 45 minutes for standard brain MRIs.
Drug: Bevacizumab — A cycle is defined as 28 days (1 month). The study duration is 12 months (12 cycles). Patients will be treated after 12 months or at the time of progression per discretion of their responsible physician.
  Other Names: Avastin®
Drug: CCNU — A cycle is defined as 28 days (1 month). The study duration is 12 months (12 cycles). Patients will be treated after 12 months or at the time of progression per discretion of their responsible physician.
  Arms: FMISO PET & MRI Group 2

SUMMARY:
In this research study, the investigators are using FMISO-PET and MRI scans to explore the delivery of bevacizumab to the blood vessels in patient's with recurrent glioblastoma before and after treatment.

Bevacizumab is approved by the U.S. Food and Drug Administration for use in patients with recurrent glioblastoma . It works by targeting a specific protein called VEGF, which plays a role in promoting the growth or spreading of tumor blood vessels. Since anti-VEGF agents also affect normal blood vessels in the brain, they can inhibit the way other drugs used in combination with bevacizumab are delivered to the tumor.

In PET scans, a radioactive substance is injected into the body. The scanning machine finds the radioactive substance, which tends to go to cancer cells. For the PET scans in this research study, the investigators are using an investigational radioactive substance called FMISO. "Investigational" means that the role of FMISO-PET scans is still being studied and that research doctors are trying to find out more about it. FMISO goes to areas with low oxygenation so parts of the tumor that do not have enough oxygen can be seen.

In addition, a vascular MRI will be used to evaluate the changes in tumor blood flow, blood volume, and how receptive blood vessels are. This scan will be performed at the same time of the FMISO-PET scan.

DETAILED DESCRIPTION:
This study does not add any additional treatment to patients with malignant glioma who are already scheduled to receive bevacizumab monotherapy. All treatment decisions will be at the discretion of the treating physician. There will be no change in the diagnosis or management of the patient based on any procedures or tests carried out as a part of this study.

If the participant chooses to take part in this research study each treatment cycle will last 28 days.

* Day 1-The participant will have the following procedures done before they can receive bevacizumab:

  * An assessment of the participant's tumor by Vascular MRI (Magnetic Resonance Imaging) and FMISO-PET scans
  * Blood pregnancy test for women of childbearing potential.
* Day 14:The participant will have the following procedures done after they receive bevacizumab:

  * An assessment of the participant's tumor by Vascular MRI (Magnetic Resonance Imaging) and FMISO-PET scans before the participant have received bevacizumab
  * Blood pregnancy test for women of childbearing potential.
* Day 28: The participant will have the following procedures done after they receive bevacizumab:

  * An assessment of the participant's tumor by Vascular MRI (Magnetic Resonance Imaging) and FMISO-PET scans after the participant has received bevacizumab
  * Blood pregnancy test for women of childbearing potential.

FMISO-PET Scans:

* The participant will have the scans performed in Charlestown, MA at the Martinos Center. The participant will be injected with two separate intravenous (IV) injections (listed below). Intravenous means a need will be injected into a vein in the participant's arm.

  * FMISO for PET scan and a contrast dye for the MRI scan
  * Drawing blood to assess the radioactivity of FMISO
* The PET scan will take approximately 60-75 minutes. The participant will receive one injection of FMISO. Following the injection of the radiotracer, blood samples will be taken from the second IV line. The tracer is given through a vein (IV) and travels through the participant's blood and collects in organs and tissues. The participant will need to wait nearby as the tracer is absorbed by the their body. This takes about 90 minutes. Then, the participant will lie on a narrow table that slides into a large tunnel-shaped scanner. The PET will pick up signals from the tracer and a computer will change the signals into 3D pictures that will be displayed on a monitor for the participant's study doctor to read.

MRI Scan:

* MRI scans will last about 60-75 minutes. This will occur at the same time as the PET scan. The participant will be injected with contrast dye twice during the MRI scan. The participant will have 3 MRI scans (prior to starting treatment, day 1 of treatment and day 14 of treatment) that would not have routinely been performed if the participant were not participating in this study.
* Blood samples will be collected during both scans in order to measure how the participant blood vessels are processing the radiotracer FMISO and how well it is being delivered to the tumor tissue.
* The participant will be assessed for side effects via clinic visit or phone call about 24 hours after each of the visits above.

Planned Follow-up: The investigators would like to call the participant every 3 months for three years after the 28 day visit to see how they are doing and if the participant is experiencing any side effects. If the participant is removed from the study due to an unacceptable side effect, the participant will be followed until it has been resolved.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed glioblastoma and evidence of recurrence. Patients with low-grade tumors who have progressed to glioblastoma are eligible.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 10 mm. See section 10 for the evaluation of measureable disease.
* Only patients for whom their neuro-oncologist has planned to give bevacizumab as monotherapy are eligible for this study
* Age > 18 years. Because no dosing or adverse event data are currently available on the use of FMISO in participants <18 years of age, children are excluded from this study but will be eligible for future pediatric trials.
* Life expectancy of greater than 3 months.
* Karnofsky performance status > 60 (see Appendix A).
* Participants must have normal organ and marrow function as defined below:

  * Leukocytes > 3,000/mcL
  * Absolute neutrophil count > 1,500/mcL
  * Platelets > 100,000/mcL
  * Total bilirubin within normal institutional limits
  * AST (SGOT)/ALT (SGPT) < 2.5 X institutional upper limit of normal
  * Creatinine within normal institutional limits or creatinine clearance > 60 mL/min/1.73 m2 for subjects with creatinine levels about institutional normal.
* Patient must be able to undergo MRI and PET scans.
* Patients must be maintained on a stable corticosteroid regimen for 5 days prior each MR-PET scan.
* The effects of FMISO on the developing human fetus are unknown. For this reason and because radiopharmaceuticals agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to temozolomide or FMISO.
* Participants who have already received anti-VEGF or experimental anti-angiogenic therapy for glioblastoma.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because FMISO is a radiopharmaceutical agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with radiopharmaceutical agents, breastfeeding should be discontinued if the mother is treated with radiopharmaceutical agents. These potential risks may also apply to other agents used in this study.
* HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with FMISO. In addition, these individuals are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Patients who are no suitable to undergo MRI or use gadolinium contrast due to:

  * Claustrophobia
  * Presence of metallic objects or implanted medical devices in body (i.e. cardiac pacemaker, aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants)
  * Sickle cell disease
  * Renal failure
  * Reduced renal function, as determined by creatinine clearance < 30 mL/min based on a serum creatinine level obtained within 28 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-02; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Gerstner, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- FMISO PET & MRI Group 1: Bevacizumab:
  * Bevacizumab will be administered at a dose of 10 mg/kg i.v. every 14 days per standard of care and the drug label. A cycle is defined as 28 days (1 month).
    -FMISO PET Scan
  * FMISO will be intravenously injected at a dose of 3.7 MBq/kg (0.1 mCi/kg) (maximum 260 MBq, 7 mCi) in < 15 mL. The IV will remain in place for injection of the gadolinium for the MRI scan. There will be one injection of FMISO in the PET protocol. Approximately 90 minutes after the injection, the PET scan will begin.
  * The PET scan will be approximately 60-75 minutes.
    -MRI
  * Each MRI will last 60-75 minutes versus 45 minutes for standard brain MRIs.
  FMISO PET
  MRI: MR scans will be performed with the same sequences and in the same order during each visit, including T1- and T2-weighted volumetric images, fluid attenuated inversion recovery (FLAIR), contrast agent enhanced T1-weighted permeability, diffusion tensor imaging (DTI), T2/T2*-weighted perfusion scans, and MR Spectroscopy. The "Autoalign" package available from the manufacturer will be used to achieve the same slice prescription in the same patient at each visit. Each MRI will last 60-75 minutes versus 45 minutes for standard brain MRIs.
  Bevacizumab: A cycle is defined as 28 days (1 month). The study duration is 12 months (12 cycles). Patients will be treated after 12 months or at the time of progression per discretion of their responsible physician.
- FMISO PET & MRI Group 2: Bevacizumab + CCNU:
  * Bevacizumab administered at dose of 10 mg/kg IV every 14 days per standard of care and drug label. Cycle defined as 28 days (1 month). Patients will be treated after 12 months or at the time of progression per discretion of their responsible physician.
  * CCNU administered at dose of 110 mg/m2 every 42 days per standard of care and drug label. Cycle defined as 28 days (1 month). Patients will be treated after 12 months or at the time of progression per discretion of their responsible physician.
    -FMISO PET Scan
  * FMISO intravenously injected at dose of 3.7 MBq/kg (0.1 mCi/kg) (maximum 260 MBq, 7 mCi) in < 15 mL. IV will remain in place for injection of gadolinium for MRI scan. One injection of FMISO in PET protocol. Approximately 90 min after injection, PET scan will begin.
  * PET scan will be approximately 60-75 minutes
    - MRI
  * Each MRI will last 60-75 minutes vs 45 minutes for standard brain MRIs.
  FMISO PET
  MRI: MR scans will be performed with the same sequences and in the same order during each visit, including T1- and T2-weighted volumetric images, fluid attenuated inversion recovery (FLAIR), contrast agent enhanced T1-weighted permeability, diffusion tensor imaging (DTI), T2/T2*-weighted perfusion scans, and MR Spectroscopy. The "Autoalign" package available from the manufacturer will be used to achieve the same slice prescription in the same patient at each visit. Each MRI will last 60-75 minutes vs 45 minutes for standard brain MRIs.
Period: Overall Study
Arm/Group | FMISO PET & MRI Group 1 | FMISO PET & MRI Group 2
Started | 2 | 9
Completed | 2 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- FMISO PET & MRI Group 1: Bevacizumab:
  * Bevacizumab will be administered at a dose of 10 mg/kg i.v. every 14 days per standard of care and the drug label. A cycle is defined as 28 days (1 month).
    -FMISO PET Scan
  * FMISO will be intravenously injected at a dose of 3.7 MBq/kg (0.1 mCi/kg) (maximum 260 MBq, 7 mCi) in < 15 mL. The IV will remain in place for injection of the gadolinium for the MRI scan. There will be one injection of FMISO in the PET protocol. Approximately 90 minutes after the injection, the PET scan will begin.
  * The PET scan will be approximately 60-75 minutes.
    - MRI
  * Each MRI will last 60-75 minutes versus 45 minutes for standard brain MRIs.
  FMISO PET
  MRI: MR scans will be performed with the same sequences and in the same order during each visit, including T1- and T2-weighted volumetric images, fluid attenuated inversion recovery (FLAIR), contrast agent enhanced T1-weighted permeability, diffusion tensor imaging (DTI), T2/T2*-weighted perfusion scans, and MR Spectroscopy. The "Autoalign" package available from the manufacturer will be used to achieve the same slice prescription in the same patient at each visit. Each MRI will last 60-75 minutes versus 45 minutes for standard brain MRIs.
  Bevacizumab: A cycle is defined as 28 days (1 month). The study duration is 12 months (12 cycles). Patients will be treated after 12 months or at the time of progression per discretion of their responsible physician.
- Total: Total of all reporting groups
Arm/Group | FMISO PET & MRI Group 1 | FMISO PET & MRI Group 2 | Total
Number analyzed (Participants) | 2 | 9 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 8 | 8
  >=65 years | 2 | 1 | 3
Age, Continuous [Median (Full Range); unit: years] | 75 [73 to 77] | 54 [29 to 70] | 58 [29 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 8 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 2 | 8 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 7 | 9
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Tumor Blood Flow/Perfusion
Description: In this research study, the investigators are using FMISO-PET and MRI scans to explore the delivery of bevacizumab to the blood vessels in patient's with recurrent glioblastoma before and after treatment.
Time Frame: Baseline and day 14 scans
Population: Group 1 (Bevacizumab monotherapy) enrolled 2 patients. Group 2 (Bevacizumab+Lomustine) enrolled 9 patients. Any analysis per arm would be meaningless so the outcome data for both groups were lumped together. There was no pre-specified analysis plan to analyze the cohorts separately. Due to production challenges with FMISO, only 4 patients underwent all 3 FMISO-PET scans: baseline, day 14, and day 28. All 4 patients were in Group 2. The remaining 7 patients had MRI scans alone at those visits.
Measure: Median (Inter-Quartile Range); unit: mL/100 g/min
Groups:
- FMISO PET & MRI (Combined Groups): Bevacizumab + CCNU:
  * Bevacizumab administered at dose of 10 mg/kg IV every 14 days per standard of care and drug label. Cycle defined as 28 days (1 month). Patients will be treated after 12 months or at the time of progression per discretion of their responsible physician.
  * CCNU administered at dose of 110 mg/m2 every 42 days per standard of care and drug label. Cycle defined as 28 days (1 month). Patients will be treated after 12 months or at the time of progression per discretion of their responsible physician.
    -FMISO PET Scan
  * FMISO intravenously injected at dose of 3.7 MBq/kg (0.1 mCi/kg) (maximum 260 MBq, 7 mCi) in < 15 mL. IV will remain in place for injection of gadolinium for MRI scan. One injection of FMISO in PET protocol. Approximately 90 min after injection, PET scan will begin.
  * PET scan will be approximately 60-75 minutes
    - MRI
  * Each MRI will last 60-75 minutes vs 45 minutes for standard brain MRIs.
  FMISO PET
  MRI: MR scans will be performed with the same sequences and in the same order during each visit, including T1- and T2-weighted volumetric images, fluid attenuated inversion recovery (FLAIR), contrast agent enhanced T1-weighted permeability, diffusion tensor imaging (DTI), T2/T2*-weighted perfusion scans, and MR Spectroscopy. The "Autoalign" package available from the manufacturer will be used to achieve the same slice prescription in the same patient at each visit. Each MRI will last 60-75 minutes vs 45 minutes for standard brain MRIs.
Arm/Group | FMISO PET & MRI (Combined Groups)
Number analyzed (Participants) | 11
mL/100 g/min
  Baseline | 1.00 [0.83 to 1.36]
  Day 14 (Week 2) | 1.15 [0.92 to 1.28]

2. Primary Outcome: Change in Tumor Hypoxic Volume
Description: In this research study, the investigators are using FMISO-PET and MRI scans to explore the delivery of bevacizumab to the blood vessels in patient's with recurrent glioblastoma before and after treatment. Regional hypoxic volume (HV) was determined by thresholding the ratio of the standardized uptake values (SUV) of FMISO in the brain to cerebellum above 1.2. Since some patients had multiple tumors, we identified the HV region within the union of each contrast enhancing region of interest (ROI) and its surrounding FLAIR ROI, so individual tumors could be evaluated separately. HV represents the magnitude of hypoxia within each tumor.
Time Frame: Baseline and day 14 scans
Population: as for outcome 1
Measure: Median (Full Range); unit: percentage of total tumor area
Arm/Group | FMISO PET & MRI (Combined Groups)
Number analyzed (Participants) | 9
percentage of total tumor area
  Baseline | 45 [40 to 74]
  Day 14 (Week 2) | 62 [43 to 88]

3. Secondary Outcome: Blood Vessel Permeability (Ktrans Change on MRI Scan)
Description: The DCE-MRI data were processed using in-house custom software written in MATLAB to obtain maps of Ktrans based on the 2-parameter Tofts model. Population-level arterial input functions (AIFs) were used for DCE analysis; DCE was used only to calculate Ktrans. Median tumor values for Ktrans were calculated from the contrast enhancing region of interest (ROI). Higher value is more permeability.
Time Frame: Baseline and day 14
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: 1/min
Arm/Group | FMISO PET & MRI (Combined Groups)
Number analyzed (Participants) | 11
1/min
  Baseline | 0.14 [0.06 to 0.26]
  Day 14 (Week 2) | 0.08 [0.03 to 0.13]

4. Secondary Outcome: Tumor Blood Flow Measured by MRI Perfusion
Description: This outcome measure looks at what blood flow was doing in tumor regions that were hypoxic. This outcome measured blood flow to the tumor using an MRI technique called dynamic susceptibility contrast enhancement that measures how fast injected contrast material flows through the tumor. This outcome specifically explored how blood flow to the tumor influenced tumor hypoxia.
Time Frame: Baseline and day 14 scans
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mL/100 g/min
Arm/Group | FMISO PET & MRI (Combined Groups)
Number analyzed (Participants) | 11
mL/100 g/min
  Baseline | 1.00 [0.83 to 1.36]
  Day 14 (Week 2) | 1.15 [0.92 to 1.28]

ADVERSE EVENTS:
Time Frame: Protocol only collected adverse events related to FMISO-PET scan, within 24 hrs (+/- 6 hrs) post-scan. FMISO-PET scans were done at baseline, day 14, and day 28 prior to administration of bevacizumab +/- lomustine.
Description: Adverse event data was systematically assessed by regular investigator assessment and laboratory testing. Protocol only collected adverse events related to FMISO-PET scan, within 24 hrs (+/- 6 hrs) post-scan.
Arm/Group | FMISO PET & MRI Group 1 | FMISO PET & MRI Group 2
All-Cause Mortality (participants affected / at risk) | 2/2 | 8/9
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/9
Other Adverse Events (participants affected / at risk) | 0/2 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/52/NCT02076152/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/52/NCT02076152/ICF_001.pdf